CLINICAL TRIAL: NCT07316036
Title: The Effect of Patterned Versus Plain Fixation Materials on Pain and Physiological Parameters in Children Receiving Intravenous Therapy: A Randomized Two-Period Crossover Trial
Brief Title: Effect of Patterned Versus Plain Fixation on Pain During IV Therapy in Children
Acronym: P-FLACC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Müberra Ahsen Kalburcu, Pediatric Nurse, Graduate Researcher, Necmettin Erbakan University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: NEU-IV-FLACC-2025
Record Dates: First submitted 2025-12-10; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2026-01

CONDITIONS: Pain; Intravenous Therapy; Kronik hastalık
Keywords: çocuklarda ağrı; desenli tespit malzemesi; non farmakolojik yöntemler; fizyolojik parametreler; ağrı puanı
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: This study uses a two-period randomized crossover design. Participants are assigned to one of two sequences (patterned fixation first, then plain; or plain fixation first, then patterned). Each child receives both interventions on different treatment days, serving as their own control.
Masking Description: No masking was applied because the intervention involved visibly different fixation materials (patterned versus plain), making blinding of participants and healthcare providers not feasible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patterned Fixation Material (Active Comparator): Children receive intravenous catheter fixation using patterned fixation materials during routine intravenous therapy.
  Interventions: Device: Patterned fixation tape; Device: Plain fixation tape
- Plain Fixation Material (Active Comparator): Children receive intravenous catheter fixation using standard plain fixation materials during routine intravenous therapy.
  Interventions: Device: Patterned fixation tape; Device: Plain fixation tape

INTERVENTIONS:
Device: Patterned fixation tape — Patterned fixation tape is applied to secure the intravenous catheter after insertion, with the patterned surface remaining visible to the child during the procedure.
Device: Plain fixation tape — Plain fixation tape is applied to secure the intravenous catheter after insertion using standard, non-patterned fixation materials.

SUMMARY:
The goal of this clinical trial is to learn whether using patterned fixation materials during intravenous therapy can reduce pain and affect physiological responses in children.

Children who regularly receive intravenous therapy will take part in this study. Each participant will receive both patterned and plain fixation materials on different treatment days. Pain levels will be measured using an observation-based pain scale, and oxygen saturation and pulse rate will be recorded before and after the procedure.

DETAILED DESCRIPTION:
This study is a randomized two-period crossover clinical trial designed to examine whether patterned fixation materials used during intravenous (IV) catheter placement reduce pain and influence physiological responses in children. The trial focuses on children who regularly receive IV therapy for chronic conditions and aims to compare two commonly used fixation materials: patterned fixation tape and plain fixation tape.

Participants are randomly assigned to one of two sequences. In Sequence AB, children receive the patterned fixation material during their first IV procedure and the plain fixation material during their next scheduled IV procedure. In Sequence BA, children receive the plain fixation material first and the patterned fixation material during their next procedure. A washout period of at least one week naturally occurs between visits because children attend the day treatment unit weekly or every three weeks for routine therapy. This interval is considered sufficient to prevent carry-over effects, as the intervention is a short-term non-pharmacological distraction method.

During each IV procedure, pain is assessed using the FLACC behavioral pain scale by two independent observers, and physiological parameters (oxygen saturation and pulse rate) are measured one minute before and one minute after the procedure. Each child serves as their own control, allowing within-participant comparisons between the patterned and plain fixation conditions.

The primary objective of the study is to determine whether patterned fixation materials lower pain scores compared with plain fixation materials. Secondary objectives include examining whether patterned fixation materials lead to more favorable physiological responses during IV catheter insertion.

ELIGIBILITY:
Inclusion Criteria:- Children aged between 3 and 12 years

* Children who regularly receive intravenous therapy for chronic conditions
* Ability of the child and parent/legal guardian to understand the study procedures
* Written informed consent obtained from the parent or legal guardian
* Assent obtained from the child when appropriate

Exclusion Criteria:

* - Presence of acute pain at the time of the procedure
* Diagnosis of conditions that may interfere with pain assessment, such as cerebral palsy or neuromuscular or peripheral nervous system disorders
* Requirement for more than one intravenous catheter insertion attempt during the procedure
* Withdrawal of consent by the child or parent/legal guardian

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-12-20 (Actual); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | Immediately after intravenous fixation during each study period
  Pain intensity was assessed using the FLACC (Face, Legs, Activity, Cry, Consolability) observational pain scale.
  The total score ranges from 0 to 10, with higher scores indicating more severe pain.

SECONDARY OUTCOMES:
Physiological parameters, Spo2 | Immediately before and immediately after each intervention period
  Oxygen saturation (SpO₂) measured before and after intravenous fixation.
Physiological parameters, heart rate | Immediately before and immediately after each intervention period
  heart rate measured before and after intravenous fixation.

CONTACTS AND LOCATIONS:
Locations (1):
- Necmettin Erbakan Üniversitesi, Konya, Meram, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared because the study involves pediatric patients and includes sensitive clinical information. The informed consent forms and ethical approval for this thesis project do not allow the sharing of identifiable or individual-level data with external researchers.